CLINICAL TRIAL: NCT06797336
Title: A Phase 1, Open-Label Dose Escalation and Expansion Study of PT0253 in Participants With KRAS G12D Mutated Advanced Solid Tumors
Brief Title: A Study of PT0253 in Participants With KRAS G12D Mutated Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PAQ Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PT0253-101
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor
Keywords: KRAS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1a, Dose Escalation (Experimental): Participants with any type of solid tumor will receive PT0253 injection, intravenously (IV) until disease progression or intolerance.
  Interventions: Drug: PT0253
- Part 1b, Dose Expansion: Tumor type 1 (Experimental): Participants with a previously treated tumor type will receive PT0253 injection until disease progression or intolerance. Recommended dose or doses for expansion for Part 1b will be determined based on the safety, tolerability, pharmacokinetic (PK) and pharmacodynamic (PD) data for PT0253 established in Part 1a.
  Interventions: Drug: PT0253
- Part 1b, Dose Expansion: Tumor type 2 (Experimental): Participants with a previously treated tumor type will receive PT0253 injection until disease progression or intolerance. Recommended dose or doses for expansion for Part 1b will be determined based on the safety, tolerability, PK and PD data for PT0253 established in Part 1a.
  Interventions: Drug: PT0253
- Part 1b, Dose Expansion: Tumor type 3 (Experimental): Participants with a previously treated tumor type will receive PT0253 injection until disease progression or intolerance. Recommended dose or doses for expansion for Part 1b will be determined based on the safety, tolerability, PK and PD data for PT0253 established in Part 1a.
  Interventions: Drug: PT0253

INTERVENTIONS:
Drug: PT0253 — PT0253 injection.

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability, determine the maximally tolerated dose (MTD) and/or recommended Phase 2 dose(s) (RP2D) of PT0253 in adult participants with Kirsten rat sarcoma viral oncogene homolog (KRAS) G12D mutated advanced solid tumors as monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced or metastatic solid malignancy
2. Participant has a pathologically documented, locally advanced or metastatic malignancy with KRAS p.G12D mutation identified through molecular testing using a validated institutional or commercial test.
3. Measurable disease (RECIST 1.1 Criteria).
4. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
5. Willingness to avoid pregnancy or fathering children from screening through 90 days after the last dose of study treatment.

Exclusion Criteria:

1. Active brain metastasis or carcinomatous meningitis. If participants have had brain metastases resected or have received radiation therapy, they may be eligible if: (1) study treatment begins at least 4 weeks from the end of brain-specific therapy, (2) residual neurological symptoms Grade less than or equal to (<=) 2, (3) currently on stable doses of corticosteroids, and (4) pre-study brain magnetic resonance imaging (MRI) documents no new/worsening brain lesions.
2. History of any other malignancy within the past 2 years, except:

   * Malignancy treated with curative intent and with no known active disease present >=2 years before enrolment and felt to be at low risk for recurrence by the investigator
   * Basal or squamous cell carcinoma of the skin, in situ cervical cancer, early -stage endometrial cancer that has been definitively treated, superficial bladder cancer, Gleason 6/7 treated prostate cancer, and ductal carcinoma in situ or lobular carcinoma in situ of the breast.
3. Unresolved toxicities from prior anti-cancer therapies (Common Terminology Criteria for Adverse Events [CTCAE] grades >1), except for alopecia. Grade <=2 toxicities from prior anti-tumor therapies that are considered irreversible may be allowed, provided that they are not described in the exclusion criteria AND the investigator and medical monitor are in agreement to proceed.
4. Concurrent participation in another interventional clinical study.
5. Treatment with anticancer medications or investigational drugs within 14-28 days or 5 half-lives (whichever is longer) before the first administration of study drug. Concurrent hormonal therapy for prostate or breast cancer is allowed.
6. Significant cardiovascular disease within 6 months of starting study therapy.
7. Active infection requiring antibiotics within 1 day of study treatment.
8. Known HIV infection with a cluster of differentiation 4+ (CD4+) T-cell count less than (<) 200 cells per microliter [/mcL] and/or a detectable viral load per parameters of assay and/or on an anti-retroviral regimen containing a strong or moderate cytochrome (CY)P3A4/5 inhibitor or inducer and/or on a new anti-retroviral regimen for less than 28 days prior to the initiation of study treatment.
9. Known history of drug-induced liver injury; primary biliary cirrhosis; or ongoing extrahepatic obstruction caused by stones, cirrhosis of the liver, or portal hypertension.
10. Major surgery within 4 weeks of the start of study therapy or postoperative complications preventing the participant from adhering to protocol assessments and procedures.
11. Known hypersensitivity to any of the products to be administered during dosing.
12. Any disease or disorder that, in the opinion of the investigator, may compromise the ability of the participant to provide written informed consent and/or to comply with all required study procedures.
13. Part 1a (Dose escalation): Use of a strong or moderate CYP3A4/5 inhibitor or inducer, strong P-glycoprotein (P-gp) inhibitor or inducer or P-gp substrate.
14. Use of multidrug and toxin extrusion protein 1 (MATE) or MATE2-K substrates that cannot be discontinued prior to the start of study treatment.
15. Participants with laboratory values indicating inadequate hematology, hepatic, or renal function.
16. Clinically significant abnormalities in rhythm, conduction, or morphology of resting electrocardiogram (ECG) or baseline QT interval corrected for heart rate using Fridericia's formula (QTcF) >=450 milliseconds (msec).
17. Female participants who are pregnant or lactating/breast feeding or who plan to breastfeed while on study through 28 days after receiving the last dose of study drug.
18. Active hepatitis B virus (HBV) infection. Participants with resolved infection or who are on stable antiviral therapy are eligible.
19. Active hepatitis C virus (HCV) infection. Participants who have completed definitive antiviral therapy with post treatment confirmation of eradication are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-06-16 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting Toxicities (DLT) | Cycle 1 (Cycle length=21 days)
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to 24 months
Number of Participants with TEAEs Leading to Treatment Interruptions, Dose Reductions and Permanent Discontinuations | Up to 24 months

SECONDARY OUTCOMES:
Cmax/C0: Maximum Blood Concentration (Cmax) and/or Concentration at Time 0 (C0) of PT0253 | Cycle 1 Days 1 and 15: Pre-infusion and up to 24 hours post-infusion (Cycle length=21 days)
Tmax: Time to Reach Cmax of PT0253 | Cycle 1 Days 1 and 15: Pre-infusion and up to 24 hours post-infusion (Cycle length=21 days)
AUC0-t: Area Under the Curve From time 0 to the time of the Last Quantifiable Concentration of PT0253 | Cycle 1 Days 1 and 15: Pre-infusion and up to 24 hours post-infusion (Cycle length=21 days)
t1/2: Terminal Elimination Half-life of PT0253 | Cycle 1 Days 1 and 15: Pre-infusion and up to 24 hours post-infusion (Cycle length=21 days)
AUC0-∞: Area Under the Curve From Time 0 Extrapolated to Infinity of PT0253 | Cycle 1 Days 1 and 15: Pre-infusion and up to 24 hours post-infusion (Cycle length=21 days)
CL: Clearance of PT0253 | Cycle 1 Days 1 and 15: Pre-infusion and up to 24 hours post-infusion (Cycle length=21 days)
Vd: Volume of Distribution of PT0253 | Cycle 1 Days 1 and 15: Pre-infusion and up to 24 hours post-infusion (Cycle length=21 days)
Overall Response Rate (ORR) | Up to 24 months
  ORR will be determined by radiographic disease assessments per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Duration of Response (DOR) | Up to 24 months
  DOR will be determined by radiographic disease assessments per RECIST 1.1.
Overall Survival (OS) | At 1 year
  OS is defined as the time from enrollment up to death due to any cause.
Progression-free Survival (PFS) | At 1 year
  PFS will be determined by radiographic disease assessments per RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Dana Farber/Massachusetts General Hospital, Inc, Boston, Massachusetts
  - SCRI Lake Mary, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - New Experimental Therapeutics of San Antonio LLC, San Antonio, Texas
  - START - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah
  - NEXT Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes